CLINICAL TRIAL: NCT00084461
Title: Phase II Study of Depsipeptide in Metastatic Neuroendocrine Tumors
Brief Title: Romidepsin in Treating Patients With Locally Advanced or Metastatic Neuroendocrine Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01449; 0425; NCI-6325; OSU-2003C0085; CDR0000365313; U01CA076576 (NIH)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Gastrinoma; Glucagonoma; Insulinoma; Metastatic Gastrointestinal Carcinoid Tumor; Pancreatic Polypeptide Tumor; Pulmonary Carcinoid Tumor; Recurrent Gastrointestinal Carcinoid Tumor; Recurrent Islet Cell Carcinoma; Regional Gastrointestinal Carcinoid Tumor; Somatostatinoma
MeSH Terms: conditions — Gastrinoma; Glucagonoma; Insulinoma; Carcinoma, Islet Cell; Somatostatinoma | interventions — romidepsin

ARMS (1):
- Treatment (romidepsin) (Experimental): Patients receive romidepsin IV over 4 hours on days 1, 8, and 15. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients achieving CR receive 2 additional courses beyond CR.
  Interventions: Drug: romidepsin; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: romidepsin — Given IV
  Other Names: FK228; FR901228; Istodax
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of romidepsin in treating patients who have locally advanced or metastatic neuroendocrine tumors. Drugs used in chemotherapy, such as romidepsin, work in different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine objective response rate in patients with locally advanced or metastatic neuroendocrine tumors treated with FR901288 (romidepsin).

SECONDARY OBJECTIVES:

I. Determine the toxicity of this drug in these patients. II. To measure serum tumor markers (pancreastatin, gastrin, pancreatic polypeptide, glucagon, substance-P, neurotensin, calcitonin, somatostatin, vasoactive intestinal peptide, gastrin releasing polypeptide, ACTH) depending on the tumor type pre-, during-, and post-treatment.

III. To perform a nuclear medicine functional imaging scan (octreoscan) to evaluate the disease status pre-, during-, and post-treatment.

IV. To perform histone acetylation assay in cytospins from peripheral blood mononuclear cells (PBMCs) to correlate with disease response and with immunologic parameters.

V. To quantify gene expression by Real Time PCR of type 1 and type 2 cytokines, co-stimulatory molecules, and adhesion molecules in PBMCs obtained from the pre-, during-, and post-treatment blood samples.

VI. To perform a multicolor flow cytometric analysis on fresh blood to assess activation of lymphocyte subsets and presence of co-stimulatory and adhesion molecules.

VII. To perform in vitro functional assays for innate as well as antigen-specific T cell immune responses in PBMCs obtained from the pre-, during-, and post-treatment blood samples.

OUTLINE:

Patients receive romidepsin IV over 4 hours on days 1, 8, and 15. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients achieving complete remission (CR) receive 2 additional courses beyond CR.

Patients are followed at 2-4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed carcinoid tumor or islet cell neuroendocrine tumor

  * Well- or moderately-differentiated tumor
* Metastatic and/or locally advanced disease
* Measurable disease

  * Unidimensionally measurable lesion at least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
  * Lesions in a previously irradiated area are not considered measurable
  * No truly non-measurable lesions, including the following:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural or pericardial effusion
    * Lymphangitis cutis/pulmonis
    * Abdominal masses not confirmed and followed by imaging
    * Cystic lesions
* Ineligible for standard treatment
* Performance status - ECOG 0-1
* At least 6 months
* WBC >= 3,000/mm^3
* Absolute neutrophil count >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Bilirubin =< 1.5 mg/dL
* AST and ALT =< 2.5 times upper limit of normal
* Creatinine =< 1.5 mg/dL
* No New York Heart Association class III or IV congestive heart failure
* No myocardial infarction within the past year
* No uncontrolled dysrhythmias
* No poorly controlled angina
* No serious ventricular arrhythmia, defined as ventricular tachycardia or ventricular fibrillation >= 3 beats in a row
* No left ventricular hypertrophy by EKG
* No other significant cardiac disease
* QTc < 500 msec
* LVEF > 40% by resting MUGA
* No prior allergic reaction attributed to compounds of similar chemical or biological composition to study drug
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No other concurrent uncontrolled illness
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* More than 4 weeks since prior immunotherapy (e.g., interferon alfa)
* More than 4 weeks since prior chemotherapy
* More than 12 weeks since prior hepatic artery chemoembolization unless liver lesions are not the only indicator lesions
* No prior FR901228 (depsipeptide)
* No more than 1 prior systemic chemotherapy regimen for carcinoid or islet cell tumor (other than hepatic artery chemoembolization)
* More than 4 weeks since prior oral or IV steroids (first 16 patients only)
* Concurrent long-acting octreotide allowed at standard doses if dose has been stable for the past 12 weeks

  * Concurrent subcutaneous octreotide for breakthrough use for symptomatic relief allowed
* No concurrent systemic steroids (first 16 patients only)
* More than 4 weeks since prior radiotherapy
* More than 4 weeks since prior investigational tumor-specific therapy
* No other prior histone deacetylase inhibitors (e.g., valproic acid)
* No concurrent hydrochlorothiazide
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational or commercial agents or therapies for the malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2004-03; Primary Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Objective response rate | Up to 4 weeks
  Frequency of response will be estimated with a 95% confidence interval.

SECONDARY OUTCOMES:
Incidence of toxicity | Up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Shah, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States